CLINICAL TRIAL: NCT06490913
Title: Chemotherapy Plus EGFR Monoclonal Antibody in Patients With Liver Metastases From Colorectal Cancer With ctDNA Superselective Negative Genes：a Phase II Single-arm Study
Brief Title: Chemotherapy Plus EGFR Monoclonal Antibody in Patients With Liver Metastases From Colorectal Cancer With ctDNA Superselective Negative Genes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-01
Record Dates: First submitted 2024-07-01; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Liver Metastases of Colorectal Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Cetuximab; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cetuximab+chemotherapy (Experimental): XELOX 1 cycle；cetuximab+chemotherapy up to 12 cycles
  Interventions: Drug: Capecitabine; Drug: oxaliplatin; Drug: Cetuximab; Drug: Leucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: Capecitabine — 1000mg/m2, bid, d1-d14，q3w，1cycle
Drug: oxaliplatin — 130mg/m2, ivgtt, d1，q3w，1cycle
Drug: Cetuximab — cetuximab 500mg/m2, q2w
Drug: Oxaliplatin — 85mg/m2, d1,q2w
Drug: Leucovorin — 400mg/m2, d1,q2w
Drug: 5-FU — 400mg/m2，d1,q2w

SUMMARY:
The purpose of this Phase II single-arm study is to prospectively explore the efficacy of chemotherapy plus EGFR inhibitors in patients with liver metastases from total wild-type colorectal cancer with ctDNA superselective negative genes.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years (including 18 and 75 years);
* ECOG PS 0 or 1;
* Colorectal cancer diagnosed histologically and/or cytologically with metastatic or recurrent lesions that are not curable with surgery;
* Patients with liver metastases of RAS wild-type colorectal cancer who have not received prior treatment;
* At least one measurable lesion as defined in RECIST version 1.1;
* Fertile patients must be willing to take highly effective pregnancy avoidance measures during the study period and ≥120 days after the last dosing; Female patients with negative urine or serum pregnancy test results within ≤7 days before the first administration of the study drug;
* Have fully understood the study and voluntarily signed the informed consent.
* Adequate organ and bone marrow function, meeting the following definitions:

  1. Blood routine (no transfusion, no use of granulocyte colony stimulating factor [G-CSF], no use of other drugs for correction within 14 days before treatment); Absolute neutrophil count (ANC) ≥1.5×109/L; Hemoglobin (HB) ≥9.0 g/dL; Platelet count (PLT) ≥80×109/L;
  2. Blood biochemistry, serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN) or creatinine clearance ≥60 mL/min; Serum albumin ≥2.8g/dL. Patients with poor nutritional status before neoadjuvant therapy could also be enrolled if they met the criteria through parenteral nutrition. Total bilirubin (TBIL) ≤ 1.5×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤2.5×ULN;

Exclusion Criteria:

* Pregnant or lactating women;
* Patients with a known history of allergy to any investigative drug, similar drug, or excipient;
* Patients with risk of massive gastrointestinal bleeding or gastrointestinal obstruction;
* Patients with a history of thromboembolism, except thrombosis caused by PICC;
* There are patients with active infection;
* Patients with difficult to control hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90mmHg);
* Patients with brain metastases with clinical symptoms or imaging evidence;
* Treatment contraindications exist in combination with other chronic diseases;
* Patients with previous immunotherapy-related myocarditis, pneumonia, colitis, hepatitis, nephritis and other conditions, and the current AE is still ≥ grade 2;
* According to NCI CTCAE version 5.0 evaluation criteria, existing patients with various toxic and side effects caused by previous treatment ≥ grade 2;
* Other conditions that the investigator determined were not suitable for inclusion in the study.
* Received any anti-tumor therapy and participated in other clinical studies within 4 weeks before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | every 2 weeks

SECONDARY OUTCOMES:
overall survival | Around 2 years